CLINICAL TRIAL: NCT01881620
Title: PET / Enhanced CT Scan Performance in Cancer (Positron Emission Tomography Combined With Computed Tomography or Vascular Contrast CT Scan). COMBI TEP Study
Brief Title: PET Enhanced CT Scan Performance in Cancer
Acronym: COMBITEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IB2009-70
Record Dates: First submitted 2012-11-05; First posted 2013-06-19 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2019-07

CONDITIONS: Cancer Disease Progression
Keywords: PET scan; CT scan; Diagnostic performance
MeSH Terms: conditions — Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COMBI TEP : PET / enhanced CT scan (Experimental): COMBI TEP : PET / enhanced CT scan
  Interventions: Device: COMBI TEP : PET / enhanced CT scan

INTERVENTIONS:
Device: COMBI TEP : PET / enhanced CT scan — diagnostic imaging exam
  Other Names: diagnostic imaging exam

SUMMARY:
Hypothesis:

The investigators would like to demonstrate that diagnosis performance of PET/CT scan without and with contrast agent (COMBI TEP), are equivalent or better than those of PET/ non enhanced CT scan (PET scan) associated with an enhanced CT scan. This research project is a pilot study given the few available data concerning this imaging exam reproducibility.

This study is a prospective single center study.

DETAILED DESCRIPTION:
Hypothesis:

We would like to demonstrate that diagnosis performance of PET/CT scan without and with contrast agent (COMBI TEP), are equivalent or better than those of PET/ non enhanced CT scan (PET scan) associated with an enhanced CT scan. This research project is a pilot study given the few available data concerning this imaging exam reproducibility. This study allows us to assess the feasibility of such a large-scale study, but also to evaluate COMBI TEP performance. From these estimates, we can then consider a comparative study to evaluate the performance of COMBI PET.

This study is a prospective single center study.

ELIGIBILITY:
Inclusion Criteria:

Any patient with a cancerous disease for which PET scan is indicated in the SOR (Standards - Options - Recommendations) FDG PET 2003 updated in 2006 must be included in the trial, in the following locations:

1. Digestive cancers

   * Colorectal cancer

     * Preoperative evaluation in local and metastatic recurrence
     * Location of recurrences, in case of ACE increase in a previously operated patient.
   * Esophageal cancer: initial staging.
   * Pancreatic cancer

     * Initial staging,
     * Differential diagnosis with chronic pancreatitis.
   * Liver cancer: differential diagnosis of liver metastases, cholangiocarcinoma and benign tumors in the case of an isolated hepatic localization.
   * Digestive Endocrine tumors: staging in case of normal pentetreotide scintigraphy.
2. Lung cancer

   * Initial staging,
   * Diagnosis of lung isolated lesion > 1 cm.
3. Head and neck cancer

   * Initial pretreatment staging,
   * Recurrence diagnosis
4. Lymphoma

   * Initial staging of Hodgkin's disease (HD), non-Hodgkin's lymphoma (NHL) and aggressive follicular lymphomas,
   * Diagnosis of minimal residual disease of HD and aggressive NHL,
   * Early assessment of treatment response.
5. Thyroid cancer: suspicion of residual disease or relapse when conventional imaging data are insufficient.
6. Ovarian cancer recurrence
7. Age ≥ 18 years.
8. Chest-abdomen-pelvis enhanced CT scan achieved within 4 weeks before enrollment (with cuts of less than 5 mm).
9. Woman of childbearing age with negative pregnancy test and / or contraception.
10. Patient with informed consent signed.
11. Patient affiliated to social security schemes.

Exclusion Criteria:

1. Iodine known allergy.
2. Diabetes, excepted if controlled (hemoglucotest ≤ 1.6 g).
3. Known renal failure (creatinine clearance <60ml/min).
4. Indications against Xenetix ®:

   * Hypersensitivity to Xenetix ® or any of the excipients,
   * History of an immediate response or delayed cutaneous reaction to Xenetix ® injection.
   * Thyrotoxicosis.
5. Pregnant or lactating women.
6. Unable to undergo medical follow up for geographical, social or psychological reasons,
7. Private of freedom patient and adult under a legal guardianship or unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-03-19 (Actual); Primary Completion 2012-07-19 (Actual); Study Completion 2015-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CAZEAU Anne Laure, MD, Study Chair — Institut Bergonié

REFERENCES:
- See also: Site internet du promoteur, l'Institut Bergonié — https://www.bergonie.fr/les-essais-cliniques/

RESULTS

PARTICIPANT FLOW:
Groups:
- COMBI TEP : PET / Enhanced CT Scan: COMBI TEP : PET / enhanced CT scan : diagnostic imaging exam First, realisation of CT scan without injection followed by a PET scan (TEPSCAN) on the same Phillips GEMINI TF PET/CT camera.
  A few minutes after the TEPSCAN, injection CT is performed (XenetiX, iodinated contrast agent 350 mg l/mL).
  The COMBI TEP exam includes the TEP and the 2 series of scans (not injected low dose and injected full dose).
Period: Overall Study
Arm/Group | COMBI TEP : PET / Enhanced CT Scan
Started | 109
Completed | 105 (Eligible patients with PET-CT scanner performed AND interpretation of 2 pairs of observors available)
Not Completed | 4
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | COMBI TEP : PET / Enhanced CT Scan
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 63
Region of Enrollment [Number; unit: participants]
  France | 109
Weight [Mean (Standard Deviation); unit: kilogram] — Population: Missing data for 7 data
  kilogram
    number analyzed (Participants) | 102
    (all) | 69.1 (15)
height [Mean (Standard Deviation); unit: centimetre] — Population: Missing data for 37 patients
  centimetre
    number analyzed (Participants) | 72
    (all) | 168.4 (9.7)
Tumor localisation [Count of Participants; unit: Participants]
  Not available | 1
  Digestive | 66
  Lung | 17
  Ear Nose and Throat | 2
  Lymphoma | 21
  Thyroid | 1
  ovarian | 1

OUTCOME MEASURES:

1. Primary Outcome: Inter-observer (B1 and B2) Reproducibility of the PET-CT by Anatomical Regions
Description: The primary endpoint was the inter-observer reproducibility of the interpretation of the combined PET / enhanced CT scan (PET-CT) by anatomical region. Reproducibility was assessed for each of the 5 anatomical regions (thorax, abdomen, pelvis, bone, nervous system). Two independant pairs (B1 and B2), each composed of one nuclear physician and one radiologist interpreted the PET-CT examination and described each of the 5 anatomical régions according to 3 modalities (Presence of suspicious lesion(s); Presence of dubious lesion(s); Absence of suspicious and dubious lesion). The inter-observer reproducibility (inter-pairs of observers) was evaluated for each anatomical region by comparing the interpretations of the two pairs, using the weighted kappa concordance coefficient [ref = Fleiss J, Levin B, Cho Paik M. Statistical methods for rates and proportions. Third ed. 2003.].Interpretation by B1 after PET-CT examination (1 month after). Interpretation by B2 at the end of the study
Time Frame: 1 year
Population: Eligible patients with PET-CT scanner performed AND interpretation of 2 pairs of observors available.
Measure: Number (95% Confidence Interval); unit: Weighted kappa concordance coefficient
Arm/Group | COMBI TEP : PET / Enhanced CT Scan
Number analyzed (Participants) | 105
Weighted kappa concordance coefficient
  Thorax region: number analyzed (Participants) | 104
  Thorax region | 0.7254 [0.6288 to 0.8220]
  Abdomen region | 0.7854 [0.6923 to 0.8784]
  Pelvis region | 0.7597 [0.6408 to 0.8787]
  Bone region | 0.6711 [0.4239 to 0.9183]
  Nervous system region | 1 [1 to 1]

2. Secondary Outcome: Inter-observer (B1 and B2) Reproducibility of the PET-CT at a Patient Level
Description: The inter-observer reproducibility of combined PET-CT interpretations has been assessed globally for each patient. Same pairs of observer (B1 and B2) than for the primary endpoint evaluation interpreted the PET-CT examination in a global way and concluded for each patient. A weighted Kappa coefficient has been calculated from an identical methodology to that described for the primary endpoint evaluation. Interpretation by B1 was performed at least 1 month and 1 week after PET-CT examination. Interpretation by B2 was performed at the end of the study
Time Frame: 1 year
Population: Reproducibility was not calculated for 1 patient because 9 area from thorax region were not assessed by the pair of observer B2.
Measure: Number (95% Confidence Interval); unit: weighted Kappa coefficient
Arm/Group | COMBI TEP : PET / Enhanced CT Scan
Number analyzed (Participants) | 104
weighted Kappa coefficient | 0.6528 [0.5194 to 0.7863]

3. Secondary Outcome: Inter-observer (N1 and B2) Reproducibility of the PET-CT by Anatomical Regions
Description: For each of the 5 anatomical régions (thorax, abdomen, pelvis, bone, nervous system), we evaluated the reproducibility between the interpretations of the PET-CT by the nuclear physician alone (N1) and the independent pair (B2) composed by one nuclear physician and one radiologist . The nuclear physician alone (N1) and the independent pair (B2) interpreted the PET-CT examination independently and described each anatomical region.The inter-observer reproducibility has been evaluated for each anatomical region by comparing the interpretations of the nuclear physician alone and that one of independent pair of nuclear physician and radiologist, using the weighted kappa concordance coefficient [ref = Fleiss J, Levin B, Cho Paik M. Statistical methods for rates and proportions. Third ed. 2003.].Interpretation by nuclear physician alone (N1) was performed within 1 week of PET-CT examination. Interpretation by B2 was performed at the end of the study
Time Frame: 1 year
Population: Interpretation by nuclear physician alone was not performed for 1 patient
Measure: Number (95% Confidence Interval); unit: Weighted kappa concordance coefficient
Arm/Group | COMBI TEP : PET / Enhanced CT Scan
Number analyzed (Participants) | 104
Weighted kappa concordance coefficient
  Thorax region: number analyzed (Participants) | 103
  Thorax region | 0.8526 [0.7733 to 0.9319]
  Abdomen region | 0.8153 [0.7118 to 0.9187]
  Pelvis region | 0.7452 [0.6020 to 0.8885]
  Bone region | 0.8722 [0.7269 to 1.0000]
  Nervous system region | 1 [1 to 1]

4. Secondary Outcome: Inter-observer (N1 and B2) Reproducibility of the PET-CT at a Patient Level
Description: The inter-observer reproducibility of combined PET-CT interpretations has been assessed globally for each patient. The nuclear physician alone (N1) and the independent pair (B2) interpreted the PET-CT examination independently in a global way and concluded for each patient. The inter-observer reproducibility has been evaluated at patient level by comparing the interpretations of the nuclear physician alone and that one of independent pair of nuclear physician and radiologist, using the weighted kappa concordance coefficient [ref = Fleiss J, Levin B, Cho Paik M. Statistical methods for rates and proportions. Third ed. 2003.]. Interpretation by nuclear physician alone (N1) was performed within 1 week of PET-CT examination. Interpretation by B2 was performed at the end of the study
Time Frame: 1 year
Population: Interpretation by nuclear physician alone was not performed for 1 patient. Interpretation by the pair of observor B2 was incomplete for 1 patient because 9 area from thorax region were not assessed.
Measure: Number (95% Confidence Interval); unit: Weighted kappa concordance coefficient
Arm/Group | COMBI TEP : PET / Enhanced CT Scan
Number analyzed (Participants) | 103
Weighted kappa concordance coefficient | 0.7859 [0.6561 to 0.9157]

5. Secondary Outcome: Intra-observer Reproducibility of Injected CT Scan by Anatomical Regions
Description: For each anatomical region, the reproducibility of the injected CT scan was evaluated. The same radiologist evaluated the two injected CT scans (CT1 and CT2) and interpreted them (Presence of suspicious lesion(s) OR presence of dubious lesion(s) OR absence of suspicious and dubious lesion). Intra-observer reproducibility was analyzed by using the individual analysis by each radiologist. A weighted Kappa concordance coefficient was calculated per anatomical region using a methodology identical to that described for the evaluation of the proncipal endpoint. Interpretation of CT1 was performed befor inclusion. Interpretation of CT2 was performed at the end of the study.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Weighted Kappa concordance coefficient
Arm/Group | COMBI TEP : PET / Enhanced CT Scan
Number analyzed (Participants) | 105
Weighted Kappa concordance coefficient
  Thorax region | 0.8141 [0.7129 to 0.9153]
  Abdomen region | 0.7991 [0.6951 to 0.9032]
  Pelvis region | 0.7947 [0.6326 to 0.9568]
  Bone region | -0.0095 [-0.0227 to 0.0037]
  Nervous system region | 1 [1 to 1]

6. Secondary Outcome: Intra-observer Reproducibility of Injected CT Scanat a Patient Level
Description: The reproducibility of the injected CT scan was evaluated globally for each patient. The same radiologist evaluated the two injected CT scans (CT1 and CT2) and interpreted them (Presence of suspicious lesion(s) OR presence of dubious lesion(s) OR absence of suspicious and dubious lesion). Intra-observer reproducibility was analyzed by using the individual analysis by each radiologist. A weighted Kappa concordance coefficient was calculated using a methodology identical to that described for the evaluation of the proncipal endpoint. Interpretation of CT1 was performed befor inclusion. Interpretation of CT2 was performed at the end of the study.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Weighted Kappa concordance coefficient
Arm/Group | COMBI TEP : PET / Enhanced CT Scan
Number analyzed (Participants) | 105
Weighted Kappa concordance coefficient | 0.7984 [0.6708 to 0.9260]

ADVERSE EVENTS:
Arm/Group | COMBI TEP : PET / Enhanced CT Scan
Serious Adverse Events (participants affected / at risk) | 0/109
Other Adverse Events (participants affected / at risk) | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No